CLINICAL TRIAL: NCT05381636
Title: Esophageal Arterial Infusion Chemotherapy Versus Systemic Intravenous Chemotherapy for Resectable Locally Advanced Esophageal Squamous Cell Carcinoma: a Prospective, Multicentre, Randomised Controlled Clinical Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Gang Wu, Chief physician, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESCC-2022-06
Record Dates: First submitted 2022-05-15; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Resectable Locally Advanced Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Systemic intravenous chemotherapy with albumin paclitaxel 125 mg / m2 for D1, D8 + cisplatin 75 mg / m2 for D1, every 3 weeks for 1 cycle
  Interventions: Drug: Systemic intravenous chemotherapy
- Study group (Experimental): esophageal arterial infusion chemotherapy
  Interventions: Procedure: Esophageal arterial infusion chemotherapy

INTERVENTIONS:
Procedure: Esophageal arterial infusion chemotherapy — Percutaneous femoral artery puncture was performed to search for feeding arterial vessels corresponding to the lesion, and chemotherapeutic drugs were directly injected into the tumor vessels via targeted blood vessels.
  Arms: Study group
Drug: Systemic intravenous chemotherapy — Albumin paclitaxel 125 mg / m2, D1, D8 + cisplatin 75 mg / m2, D1, every 3 weeks for 1 cycle
  Arms: Control group

SUMMARY:
This was a prospective, multicentre, randomised controlled clinical study to explore the safety and efficacy of esophageal arterial infusion chemotherapy in patients with resectable locally advanced oesophageal cancer, and to compare its safety and efficacy with systemic intravenous chemotherapy. The rate of surgical R0 resection as well as progression free survival (PFS) were the main indicators.

ELIGIBILITY:
Inclusion Criteria:

* 1. Sign written informed consent prior to the implementation of any test related procedures; 2. Aged 18-75 years; 3. Histopathological examination confirmed resectable esophageal carcinoma (histologically, squamous cell carcinoma), without esophageal/gastric junction adenocarcinoma; 4. Before surgery, CT/MRI, color ultrasound, PET-CT, and ultrasonic gastroscopy were used to clearly diagnose esophageal cancer staging as >= CT3 or >=N+; 5. Newly diagnosed patients without previous surgery, radiotherapy or chemotherapy, targeted therapy or immunotherapy; 6. ECOG score ≤2，KPS ≥60%; 7. No serious heart, lung or liver dysfunction; No acute infection was associated; 8. No participation in other clinical studies within 3 months prior to treatment; 9. Sufficient organ function, subject should meet the following laboratory criteria:

  1. The absolute value of neutrophils (ANC) ≥1.5x10^9/L in the last 14 days without the use of granulocyte colony-stimulating factor;
  2. Platelets ≥80x10^9/L in the case of no blood transfusion in the last 14 days;
  3. Hemoglobin ≥80g/dL in the absence of blood transfusion or use of erythropoietin in the last 14 days;
  4. Total bilirubin ≤1.5 ULN; Or total bilirubin >ULN but direct bilirubin ≤ULN;
  5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 ULN (ALT or AST≤5 ULN are allowed in patients with liver metastasis);
  6. Serum creatinine ≤1.5 ULN and creatinine clearance rate (calculated by Cockcroft-Gault formula) ≥60ml/min;
  7. Good coagulation function, defined as INR or prothrombin time (PT) ≤1.5 ULN;
  8. Normal thyroid function is defined as thyroid stimulating hormone (TSH) within the normal range. If baseline TSH is beyond the normal range, subjects whose total T3 (or FT3) and FT4 are within the normal range can be included;
  9. Myocardial enzyme spectrum is within the normal range (if the researcher comprehensively judged that it is a simple laboratory abnormality without clinical significance, it is also allowed to be enrolled); 10. For female subjects of reproductive age, a urine or serum pregnancy test with negative results should be performed within 3 days prior to receiving the first study drug administration (cycle 1 day 1). If a urine pregnancy test cannot be confirmed negative, a blood pregnancy test is required. Women of non-reproductive age were defined as at least 1 year postmenopausal or having undergone surgical sterilization or hysterectomy; If there is a risk of conception, all subjects (both men and women) should use contraceptives with an annual failure rate of less than 1% throughout the treatment period and up to 1 year after the last study dosing.

Exclusion Criteria:

* 1. Previous operation history of thoracic malignant tumor; 2. Pathologically small cell carcinoma or distant metastasis; Patients with tumor involvement of the cervical esophagus or high upper thoracic segment requiring laryngectomy; 3. Patients with hypertension who cannot be reduced to the normal range after antihypertensive drug treatment (systolic blood pressure >140 mmHg, diastolic blood pressure > 90 mmHg); 4. Patients at high risk of bleeding or perforation due to tumor invasion of an adjacent organ of the esophageal lesion (aorta or trachea), or patients with fistula; 5. Other malignant diseases other than esophageal cancer diagnosed within 5 years prior to initial administration (excluding basal cell carcinoma of the skin after radical resection, squamous carcinoma of the skin, and/or carcinoma in situ after radical resection); 6. Is currently participating in an interventional clinical study, or has received other investigational drugs or used investigational devices within 4 weeks prior to the first administration; 7. Received Chinese patent drugs with anti-tumor indications or immunoregulatory drugs (including thymopeptide, interferon and interleukin, except for local use of pleural effusion control) within 2 weeks before the first administration; 8. Known interstitial pulmonary disease requiring steroid therapy, active pulmonary tuberculosis, active autoimmune disease requiring systemic therapy (e.g., use of palliative drugs, glucocorticoids, or immunosuppressants) developed within 2 years prior to initial administration. Alternative therapies (such as thyroxine, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic treatment; 9. The study was receiving systemic glucocorticoid therapy (excluding topical glucocorticoids by nasal spray, inhalation or other means) or any other form of immunosuppressive therapy within 7 days prior to initial administration; Note: Physiological dose of glucocorticoids (≤10mg/ day of prednisone or equivalent drug) is allowed; 10. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation; 11. People who are known to be allergic to the active ingredients or exciphers of the drugs in this study, such as cisplatin, cisplatin, or albu-paclitaxel; 12. A known history of human immunodeficiency virus (HIV) infection (i.e., HIV1/2 antibody positive); 13. The presence of any serious or uncontrollable systemic disease, such as:

  1. There are significant abnormalities in rhythm, conduction or morphology of the resting electrocardiogram with serious symptoms that are difficult to control, such as complete left bundle branch block, heart block above II degree, ventricular arrhythmia or atrial fibrillation;
  2. Unstable angina pectoris, congestive heart failure, New York Heart Association (NYHA) grade ≥2 chronic heart failure;
  3. Any arterial thrombosis, embolism or ischemia, such as myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack, occurred within 6 months before inclusion;
  4. A history of non-infectious pneumonia requiring glucocorticoid therapy or current clinically active interstitial lung disease within 1 year prior to initial administration;
  5. active tuberculosis;
  6. the presence of active or uncontrolled infections requiring systemic treatment;
  7. Clinical active diverticulitis, abdominal abscess and gastrointestinal obstruction;
  8. Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
  9. Poor control of diabetes mellitus (FBG > 14mmol/L);
  10. Routine urine indicated urinary protein ≥++, and confirmed 24-hour urinary protein quantitative > 1.0g;
  11. Patients with mental disorders who are unable to cooperate with treatment; Medical history or evidence of disease that may interfere with the outcome of the study, prevent participants from participating in the study, abnormal therapeutic or laboratory test values, or other conditions that the investigator considers unsuitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Surgical R0 resection rate | up to 1 year
Progression free survival (PFS) | up to 1 year
  PFS was defined as the time from recruitment to the first documented progressive disease (PD) or death due to any cause, whichever occurred first.

SECONDARY OUTCOMES:
Pathological complete response rate(PCRR) | up to 1 year
Objective response rate(ORR) | up to 1 year
  ORR is defined as the percentages of patients, relative to the total of enrolled subjects, achieving a complete (CR) or partial (PR) response, according to RECIST 1.1 criteria.
Treatment related AES | up to 1 year
Overall survival (OS) | up to 1 year
  The time from recruitment to death due to any cause.

IPD SHARING:
Plan to Share IPD: No